CLINICAL TRIAL: NCT02090504
Title: The Gamma Hydroxybutyric Acid in Alcohol-dependence Treatment Efficacy (GATE) I Trial: a Comparative Study Versus Oxazepam in the Treatment of Alcohol Withdrawal Syndrome
Brief Title: Comparative Study of Gamma-hydroxy Butyrate Versus Oxazepam in the Treatment of Alcohol Withdrawal Syndrome
Acronym: GATE I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: CT Pharmaceutical Industries, Sanremo - Italy (Unknown); University of Bologna (Other); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Giovanni Addolorato, Professor of Internal Medicine, Catholic University, Italy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GATE-I
Record Dates: First submitted 2014-03-17; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Alcohol Withdrawal Syndrome; Alcohol Dependence
Keywords: alcohol withdrawal syndrome; treatment; sodium oxybate; oxazepam
MeSH Terms: conditions — Alcoholism | interventions — Sodium Oxybate; Oxazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium oxybate (SMO) (Experimental): Patients randomized to the first arm of the study will receive:
  * SMO (sodium oxybate 175 mg/ml suspension): 10ml at 8.00 a.m., 10ml at 12.00 p.m., 10ml at 7.00 p.m. from day 1 to day 5, 5ml at 8.00 a.m., 5ml at 12.00 p.m., 5ml at 7.00 pm, on days 6 and 7, and 2.5ml at 8.00 a.m., 2.5 ml at 12.00 p.m., 2.5ml at 7.00 p.m. from day 8 to day 10 (If patient's weight is > 75 kg the dosage will be of 12ml instead of 10 ml, 6ml instead of 5ml, 3 ml instead of 2.5ml);
  * placebo (tablets): 1 tablet at 8.00 a.m., 1 tablet at 12.00 p.m., 1 tablet at 7.00 p.m. from day 1 to day 10.
  Interventions: Drug: Sodium Oxybate (SMO)
- Oxazepam (Active Comparator): Patients randomized to the second arm of the study will receive:
  * OXAZEPAM (tablets): 60mg at 8.00 a.m., 60mg at 12.00 p.m., 90mg at 7.00 p.m. from day 1 to day 5, 30mg at 8.00 a.m., 30mg at 12.00 p.m., 30mg at 7.00 pm, on days 6 and 7, and 15mg at 8.00 a.m., 15mg at 12.00 p.m., 15mg at 7.00 p.m. from day 8 to day 10;
  * placebo (suspension): 10ml at 8.00 a.m., 10ml at 12.00 p.m., 10ml at 7.00 p.m. from day 1 to day 5, 5ml at 8.00 a.m., 5ml at 12.00 p.m., 5ml at 7.00 pm, on days 6 and 7, and 2.5ml at 8.00 a.m., 2.5 ml at 12.00 p.m., 2.5ml at 7.00 p.m. from day 8 to day 10, (If patient's weight is > 75 kg the dosage will be of 12ml instead of 10 ml, 6ml instead of 5ml, 3 ml instead of 2.5ml).
  Interventions: Drug: Oxazepam

INTERVENTIONS:
Drug: Sodium Oxybate (SMO)
  Other Names: Gamma-hydroxy butyrate (GHB)
  Arms: Sodium oxybate (SMO)
Drug: Oxazepam
  Arms: Oxazepam

SUMMARY:
Benzodiazepines (BDZs) are the gold standard in the treatment of alcohol withdrawal syndrome (AWS). Gamma-Hydroxybutyric acid also known as sodium oxybate (SMO) has been tested as a treatment for AWS with encouraging results. Aim of this phase IV, multicenter randomized double-blind, double dummy study is to evaluate the efficacy of SMO in comparison to oxazepam in the treatment of alcohol withdrawal symptoms (AWS).

DETAILED DESCRIPTION:
This is a phase IV, multicenter randomized (1:1), active drug-controlled study (double-blind, double dummy) with parallel groups evaluating the efficacy of SMO versus oxazepam in the treatment of AWS in alcohol-dependent patients.

A placebo-controlled design was considered but excluded, given that a gold standard treatment for AWS is available (i.e., BDZs).

Furthermore, considering that SMO and oxazepam have two different pharmaceutical formulation (suspension and tablets, respectively), a double-dummy design was adopted.

Thus, all subjects will receive both medications, tablets (oxazepam or placebo) and suspension (SMO or placebo), at the same time.

ELIGIBILITY:
Inclusion Criteria:

* age range 21-75,
* diagnosis of alcohol dependence according to DSM-IV criteria
* the presence of AWS as assessed by Clinical Institute Withdrawal Assessment for Alcohol-revised (CIWA-Ar) scale, a scoring system for quantitative evaluation of physical symptoms of AWS.20 Only subjects with a CIWA-Ar score equal to or higher than 10 (defined as moderate or severe AWS requiring pharmacological treatment) were ultimately enrolled in the study.

Exclusion criteria:

* ≤55 kg of body weight;
* history of withdrawal fits within 24 hours pre-study;
* history of epilepsy or epileptics seizures not properly controlled by established anti-epileptic treatment;
* dependence from narcotics, BDZs or other drugs of abuse;
* documented pre-existent hypersensitivity to SMO or to BDZs,
* renal failure (blood creatinine >2•5 mg/dl and/or documented proteinuria >500 mg/die),
* heart failure,
* severe respiratory failure
* hepatic encephalopathy stage II-IV;
* psychiatric disorders requiring treatment with psychoactive medications before the start of the study;
* treatment with clonidine, haloperidol, bromocriptine during the last 3 months prior to participation in the study;
* participation to other clinical investigations in the previous month prior to recruitment;
* females whose could not assure not to become pregnant during the 1 month period of treatment, and during the subsequent 3 weeks;
* subjects without a stable social condition or homeless.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2002-02; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of GHB compared to oxazepam on alcohol withdrawal symptoms | day 1, day 10, day 20
  The primary outcome was the reduction of symptoms of AWS reflected by the course of the total CIWA-Ar scores from the start (baseline) to the end of the study (day 10) and to the end of follow up (day 20, 10 days after drugs discontinuation).

SECONDARY OUTCOMES:
Course of alcohol abstinence | day 1, day 10, day 20
  Secondary outcome variables included the course of alcohol abstinence. In order to confirm daily alcohol abstinence, a breath analyzer was used. In addition, to define those subjects remaining abstinent throughout the whole treatment period, carbohydrate-deficient transferrin (%CDT) was evaluated at the time of screening and at the end of the treatment period.

OTHER OUTCOMES:
Craving for study drug. | day 1, day 10, day 20
  Assessment of craving for the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Otto Lesch, MD, Prof., Principal Investigator — Department of Psychiatry, University of Wien; Giovanni Addolorato, MD, Study Director — Department of Internal Medicine, Catholic University of Rome
Locations (3):
- University of Wien, Vienna, AT, Austria
- Italy (2):
  - "G. Fontana" Centre for the Study and Multidisciplinary Treatment of Alcohol Addiction, Department of Clinical Medicine, University of Bologna, Bologna, BO
  - Catholic University of Rome, Rome, Rm

REFERENCES:
- [Background] Skala K, Caputo F, Mirijello A, Vassallo G, Antonelli M, Ferrulli A, Walter H, Lesch O, Addolorato G. Sodium oxybate in the treatment of alcohol dependence: from the alcohol withdrawal syndrome to the alcohol relapse prevention. Expert Opin Pharmacother. 2014 Feb;15(2):245-57. doi: 10.1517/14656566.2014.863278. Epub 2013 Nov 28. PMID 24283802
- [Derived] Caputo F, Skala K, Mirijello A, Ferrulli A, Walter H, Lesch O, Addolorato G. Sodium oxybate in the treatment of alcohol withdrawal syndrome: a randomized double-blind comparative study versus oxazepam. The GATE 1 trial. CNS Drugs. 2014 Aug;28(8):743-52. doi: 10.1007/s40263-014-0183-1. PMID 24996524